CLINICAL TRIAL: NCT07191457
Title: In Vivo Testing: A Two-Arm, Randomized, Controlled, Investigator/Assessor-Blinded, Comparative Study to Evaluate the Safety and Efficacy of a Head Lice Physically Acting Product: ELIMAX GREEN LOTION EMOGREEN (X92001752) vs Walgreens Lice Killing Shampoo (Piperonyl Butoxide (4%),Pyrethrum Extract (Equivalent to 0.33% Pyrethrins)) in Subjects With Head Lice.
Brief Title: Safety and Efficacy of Head-lice Treatments Elimax Green Lotion and Walgreens Lice Killing Shampoo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oystershell NV (Industry)
Collaborators: Lice Solutions Resource Network (LSRN) Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OYS011-0025
Record Dates: First submitted 2025-09-02; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Head Lice
Keywords: Head Lice; Walgreens Lice Killing Shampoo; Elimax Green Lotion Emogreen; RID Super Max Solution; Pyrethrum

STUDY DESIGN:
Intervention Model Description: A Two-Arm, Randomized, Controlled, Investigator/Assessor-Blinded Comparative Study.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment with Elimax Green Lotion with Emogreen (Experimental): Lice treatment with Elimax Green Lotion (Emogreen)
  Interventions: Device: Elimax Green Lotion with Emogreen
- Treatment with Walgreens Lice Killing Shampoo (Active Comparator): Topical lice treatment with Walgreens Lice Killing Shampoo
  Interventions: Drug: Walgreens Lice Killing Shampoo

INTERVENTIONS:
Device: Elimax Green Lotion with Emogreen — STEP 1:
  Apply the lotion to dry hair, completely saturating hair and scalp. Use a towel to cover eyes and exposed skin areas. Massage from the roots to the tips, paying particular attention to the area behind the ears and the hairline at the back of the head. Leave the lotion in the hair for 10 minutes (no longer). In the case of long hair, pin the hair up away from the skin after application.
  STEP 2:
  Wash out by applying shampoo to the hair and rinsing thoroughly. Repeat if needed to fully rinse out the lotion.
  STEP 3:
  Comb to remove lice and nits. Part the hair into sections and comb one section at a time. Place the teeth of the comb as close as possible to the scalp and comb away from the scalp to the end of the hair. Use clips to pin back each section of combed hair. Clean the comb during use by wiping onto a tissue. Discard the tissue into a sealable bag. Discard the sealed bag.
  Check hair for the following 7 to 10 days. If lice or nits are present, repeat steps 1-3.
  Arms: Treatment with Elimax Green Lotion with Emogreen
Drug: Walgreens Lice Killing Shampoo — Apply thoroughly to dry hair or other affected area. For head lice, first apply behind ears and to back of neck Allow product to remain for 10 minutes, but no longer Use warm water to form a lather, shampoo, then thoroughly rinse For head lice, towel dry hair and comb out tangles Remove lice and their eggs (nits) Use a fine-tooth or special lice/nit comb. Remove any remaining nits by hand (using a throw-away glove) Hair should remain slightly damp while removing nits If hair dries during combing, dampen slightly with water For head lice, part hair into sections. Do one section at a time starting at the top of the head. Longer hair may take 1 to 2 hours. Lift a 1- to 2- inch wide strand of the hair. Place comb as close as possible to the scalp and comb with a firm, even motion away from the scalp.
  Pin back each strand of the hair after combing Clean comb often. Wipe away nits with tissue and discard in a plastic bag. Seal bag and discard bag to prevent lice from coming back.
  Arms: Treatment with Walgreens Lice Killing Shampoo

SUMMARY:
Compare efficacy and safety of Elimax Green Lotion Emogreen (RID SUper Max Solution) to that of Walgreens Lice Killing Shampoo against headlice in infested individuals. Involved subjects aged 6 months and older, of both genders, with a confirmed diagnosis of head lice infestation are included. Local and global tolerability, skin and eye irritation are monitored throughout the study. Any adverse events will be monitored and recorded.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate and compare efficacy and safety of X92001752 Emogreen with Walgreens Lice Killing Shampoo (Piperonyl Butoxide (4%), Pyrethrum Extract (Equivalent to 0.33% Pyrethrins)) against head lice (Pediculus capitis) in infested individuals. More specifically, the present study aims to confirm the clinical performance and safety of head lice treatment product: Elimax Green Lotion with Emogreen L15® (INCI C15-19 alkane) as main ingredient (X92001752). This product works in the same way as Elimax Green Lotion with Hemisqualane® (INCI hydrogenated farnesene) namely, by physically suffocating and dehydrating lice and their nits due to the presence of a bio-alkane and beeswax. They are generally combined with a lice comb in a procedure pack. Elimax Green Lotion is classified as Class I medical devices in Europe. In the US, the products are packaged with a lice comb and registered as a Lice Removal Kit, in accordance with 21 CFR 880.5960, which is 510(k)-exempt.

In line with US regulations, the guidelines for clinical trials of medical devices must be adhered to. The study will involve subjects aged 6 months and older, of both genders, with a confirmed diagnosis of head lice infestation. To support safety assessments, local and global tolerability, skin and ocular irritation, and adverse events (AEs) will be monitored and recorded.

ELIGIBILITY:
Inclusion Criteria:

* Gender: male / female.
* Female subjects with childbearing potential who test negative for pregnancy and agree to use a reliable method of birth control (as described in section7.8) or remain
* Age ≥ 6 months of age at the time of enrollment.
* Subject must have an active head lice infestation defined as at least 5 live lice (adults and/or nymphs) and 5 live nits based on magnified observations, present on the scalp and/or hair, as determined by a trained evaluator.
* Subject is in good general health based on medical history.
* Following application per designated product timeline shampoo hair using Johnson's baby shampoo (See figure 4 for shampoo image) to rinse out the product according to the study product its IFU. Subject agrees not to additionally shampoo, wash, or rinse their hair or scalp for 24-hours post treatment.
* The subject agrees not to cut or chemically treat their hair while participating in the study.
* Subject agrees to follow all study instructions, including attending all follow-up appointments.
* Agree to not use any other anti-lice treatment or medicated hair grooming products for the duration of the study (through Day 10 visit).
* The parent or legal guardian of a child must be willing to have other family members screened for head lice. If other household members are found to have head lice and are eligible, they must be either enrolled in the study OR receive the standard of care at the site and in the same manner as study participants.
* Have a single place of residence or agree to remain at the current residence for the duration of the study.
* The subject or his/her parent/legal guardian (from age 12-17), must give written informed consent, after having been informed orally and by written text about the benefits and potential risks of the trial, as well as information regarding the insurance, taken out to cover the subjects participating in the study. A caregiver must sign an informed consent agreement for children not old enough to do so. Children aged 6-11 years of age will be administered a child's assent form. Subject or his/her parent/legal guardian must be capable of understanding and providing written informed consent.

Exclusion Criteria:

* Application of any form of head lice treatment, whether prescription or over-thecounter (OTC), or home remedy for 14 days prior to their screening visit (Visit
* Application of any topical medication of any kind on the hair or scalp for a period of 48 hours prior to the screening visit.
* Use of systemic or topical drugs or medications, including systemic antibiotics, which in the opinion of the investigative personnel may interfere with the study results.
* Known skin allergies, multiple drug allergies or multiple allergies to cosmetic products.
* History of allergy or hypersensitivity to active ingredients, or constituents of the test products.
* Subject with any visible skin/scalp condition at the treatment site which, in the opinion of the investigative personnel, will interfere with the evaluation of the test product.
* Subjects with chronic scalp disorder.
* Subject or his/her legal guardian who, in the opinion of the investigative personnel, do not understand the subject requirements for study participations and/or may be likely to exhibit poor compliance with the required visits.
* Females who are pregnant or nursing.
* Hair longer than waist length.
* Subject suspected or known not to follow instructions
* Previous participation in this study or participation in any other investigational trial within the preceding 14 days.
* The subject is directly affiliated to the investigator site personnel and/or their immediate families. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.
* The subject is an Oystershell employee or is an employee of a third-party organizations involved in the study.
* Exclude families with 4 or more household members.
* People with dreadlocks or clip in hair that cannot be removed or a person who does not want to remove these.
* Hair that is too difficult to work with, assessed by the study staff.
* Families excluded where lice exist however family member declines enrollment in the study.
* Subjects who are receiving, or are expected to receive, any antibiotic therapy during the study period will be excluded.
* No more than one working subject per household may be excluded from evaluation if he is assessed as being lice by himself or caregiver. Only working male can be excluded from evaluation if individual is bald or hair no longer than half inch and deemed lice free by himself or another adult.
* All household members of the subject, other than excluded male adult, must be screened for head lice by a licenced head lice professional. If additional household members are found to have head lice and meet the study criteria, they will be referred to LSRN Research and enrolled in study. If a household member declines enrollment, all family members will be excluded from the study.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2025-10-02 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Cure rate | From enrolment to the end of treatment on day 10
  Demonstrate that local application of Elimax Green Lotion with Emogreen achieves a cure rate that is non-inferior to Wallgreens Lice Killings Shampoo, at the end of day 10, corrected for re-infestation. A non-inferiority margin of 3% will be applied.
  If non-inferiority is established, a subsequent test will be conducted to assess whether the test product is superior to the reference product. This implies that the lower bound of the confidence interval for the difference in cure rates lies above zero.

SECONDARY OUTCOMES:
Efficacy for mild and moderate baseline infestations | From enrolment to the end of treatment on day 10
  Determine efficacy of the investigational product for head lice for mild and moderate baseline infestations (cure rate at the end of the study day 10, uncorrected as well as corrected for re-infestation).
Efficacy of the investigational product for all baseline infestations | From enrolment to the end of treatment on day 1
  Determine efficacy of the investigational product for all baseline infestations (cure rate at day 1).
Efficacy of the investigational product for mild and moderate baseline infestations. | From enrolment to the end of treatment on day 1
  Determine efficacy of the investigational product for mild and moderate baseline infestations (cure rate at day 1).
Local tolerability | From enrolment to the end of treatment on day 10
  To evaluate local tolerability by subject: subjective symptoms (burning, paraesthesia, pruritus): 0h, 1h, 24h, 7d and 10d p.a. (descriptive evaluation).
  The following 4-category scale will be used:
  * Score 1 - None: No sensation reported.
  * Score 2 - Mild: Slight, brief sensation (e.g. tingling or slight itch) easily tolerated and does not interfere with daily activities.
  * Score 3 - Moderate: Apparent discomfort (e.g. burning sensation, moderate itching) that may periodically distract or cause a minor disruption but does not require any treatment.
  * Score 4 - Severe: Prolonged or intense sensation (e.g. strong burning and/or itching) that interferes with normal activities or requires an intervention (e.g. cold compress, medication).
Global tolerability | From enrolment to the end of treatment on day 10
  Global tolerability (general well-being and global tolerability of the test product) will be assessed by the blinded study staff at day 10. The global tolerability will be rated on a 4-category scale with: Score 1 = very good, Score 2 = good, Score 3 = moderate, Score 4 = poor. Evaluation at 10d after application.
Skin irritation | From enrolment to the end of treatment on day 10
  To evaluate skin irritation by study staff (secondary infection, erythema, excoriation) on day 0, 1, 7 and 10.
  The following 4-category scale will be used:
  * Score 1 - None: No visible skin reaction.
  * Score 2 - Mild: Slight redness or dryness; with no swelling, peeling, or open sores; does not interfere with daily activities.
  * Score 3 - Moderate: Pronounced erythema, itching, or localized excoriation; may be associated with discomfort or require a non-prescription topical treatment.
  * Score 4 - Severe: Intense noticeable redness, edema, raw and/or broken skin (e.g. breakdown of skin with oozing or bleeding); may require medical intervention or lead to the discontinuation of the investigational product
Eye irritation | From enrolment to the end of treatment on day 10
  To evaluate eye irritation by study staff on day 0, 1, 7 and 10.
  The following 4-category scale will be used:
  * Score 1 - None: No redness or irritation; the eyes appear normal.
  * Score 2 - Mild: Slight conjunctival redness or dryness; with no tearing or discomfort.
  * Score 3 - Moderate: Noticeable redness with possible tearing or discomfort; does not impair vision or require any treatment.
  * Score 4 - Severe: Apparent redness with significant irritation, tearing, or pain; possibly interferes with vision or requires medical treatment.
Adverse events | From enrolment to the end of treatment on day 10
  To evaluate characterization of safety and tolerability of the investigational product considering adverse events in the study population.
Esthetical properties | The questioning will be performed on day 0 and day 7 after treatment and drying the hair.
  The esthetical properties of the investigational products will be evaluated to determine the satisfaction by the subjects with the products after application using a questionnaire about hair and scalp feeling, greasiness, hair look, shininess, and volume.
  With each question being scored on a scale from 1-4:
  * Score 1 = Strongly agree
  * Score 2 = Agree
  * Score 3 = Disagree
  * Score 4 = Strongly disagree

CONTACTS AND LOCATIONS:
Locations (1):
- LSRN Research, Enid, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No